CLINICAL TRIAL: NCT06812910
Title: Clinical Characterization and Cross-Sectional Comparison of Stigma, Mental Health, and Treatment Experience Among People Living with HIV in Urban and Insular Settings in Portugal
Brief Title: Urban and Insular Study on Treatment Experiences and Stigma in People Living with HIV
Acronym: SUNRISE
Status: Not yet recruiting | Type: Observational
Sponsor: Fábio Cota Medeiros (Network)
Responsible Party: Sponsor-Investigator, Fábio Cota Medeiros, Principal Investigator, Lisbon Academic Medical Center - Centro Académico de Medicina de Lisboa
Organization: Lisbon Academic Medical Center - Centro Académico de Medicina de Lisboa (Network)
Other Study IDs: SUNRISE
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: HIV; Stigma; Depression/Anxiety
Keywords: HIV; HIV related stigma; mental health; pill burden; treatment experience
MeSH Terms: conditions — Social Stigma; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Urban Cohort: People living with HIV (PLWH) who receive care in urban centers.
- Island Cohort: People living with HIV (PLWH) who receive care in island regions (Azores and Madeira).

SUMMARY:
Study Title: SUNRISE Study: Urban and Island Experiences of HIV Treatment and Stigma

What is this study about? This study aims to understand how living in urban areas versus islands affects the experiences of people living with HIV (PLWH) in Portugal. Specifically, the investigators want to explore how stigma and mental health (such as depression and anxiety) differ between these two settings. The investigators are also interested in understanding how the number of pills a person takes daily (called "pill burden") impacts their mental health and satisfaction with treatment.

Why is this study important? Stigma related to HIV can make it harder for people to stick to their treatment and can negatively affect their mental health and overall well-being. By comparing urban and island settings, the investigators hope to identify unique challenges faced by PLWH in different environments. This information will help the investigators to develop better strategies to support people living with HIV, no matter where they live.

Who can participate? Adults (18 years or older) who have been diagnosed with HIV. People who have been on antiretroviral therapy (HIV treatment) for at least six months.

Individuals living in urban areas or island region.

What will happen during the study?

Participants will complete a one-time interview during their regular HIV care visit. The interview will include questions about:

Their experiences with HIV-related stigma. Their mental health (including depression and anxiety). Their satisfaction with their current HIV treatment. The number of pills they take daily and how this affects their daily life. All information will be kept confidential, and participation is voluntary.

What are the potential benefits of participating? This study will help to understand the challenges faced by people living with HIV in different parts of Portugal. This knowledge can lead to improved support services and treatment options for PLWH in the future.

What are the risks of participating? There are no physical risks associated with this study. However, some questions may touch on sensitive topics, such as stigma or mental health.

How will the results be used? The results of this study will be shared with the scientific community, healthcare providers, and organizations that support people living with HIV. The goal is to use this information to improve care and reduce stigma for PLWH in Portugal and beyond.

Who is conducting this study? This study is led by researchers from the Faculty of Medicine of Lisbon, in collaboration with hospitals in Portugal mainland, the Azores, and Madeira.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with HIV
* Aged 18 years or older.
* On antiretroviral therapy (ART) for at least six months.
* On a daily oral treatment regimen (single or multiple pills).
* Able to provide informed consent.

Exclusion Criteria:

* Individuals under 18 years of age.
* Individuals who have switched antiretroviral regimen in the previous six months.
* Individuals unable to provide informed consent (e.g., due to cognitive impairment or lack of capacity).
* Individuals with limited understanding of the study procedures or questionnaires (e.g., language barriers or cognitive limitations).
* Individuals who are incarcerated or deprived of liberty.
* Pregnant individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals living with HIV (PLWH) who are receiving care in urban and island settings in Portugal. Participants must be 18 years of age or older, diagnosed with HIV, and on antiretroviral therapy (ART) for at least six months. They must also be on a daily oral treatment regimen (single or multiple pills) and able to provide informed consent.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Levels of HIV-Related Stigma in Urban versus Island Settings | Cross-sectional assessment at baseline (one-time measurement during study enrollment).
  This outcome measures the levels of HIV-related stigma experienced by individuals living with HIV (PLWH) in urban and island settings in Portugal. Stigma is assessed using a validated HIV Stigma Scale, which evaluates perceived and internalized stigma (range: 0-48, where higher scores indicate greater perceived stigma). The results will be compared between the two geographic cohorts to identify differences in stigma experiences.

SECONDARY OUTCOMES:
Prevalence of Depression and Anxiety in Urban versus Island PLWH | Cross-sectional assessment at baseline (one-time measurement during study enrollment).
  This outcome measures the prevalence of depression and anxiety among individuals living with HIV in urban and island settings. Depression is assessed using the Patient Health Questionnaire-9 (PHQ-9 ; range: 0-27, where higher scores indicate more severe depression), and anxiety is assessed using the Generalized Anxiety Disorder-7 scale (GAD-7; range: 0-21, where higher scores indicate more severe anxiety). Results will be compared between the two cohorts to identify differences in mental health outcomes.
Association Between Stigma and Mental Health Indicators (Depression and Anxiety) | Cross-sectional assessment at baseline (one-time measurement during study enrollment).
  This outcome evaluates the association between HIV-related stigma (measured using the HIV Stigma Scale; range: 0-48, where higher scores indicate greater stigma) and mental health indicators (depression measured using the Patient Health Questionnaire-9, PHQ-9; range: 0-27, where higher scores indicate more severe depression; and anxiety measured using the Generalized Anxiety Disorder-7, GAD-7; range: 0-21, where higher scores indicate more severe anxiety). The goal is to determine whether higher levels of stigma are associated with worse mental health outcomes, adjusting for potential confounding variables such as age, gender, and duration of HIV treatment. Statistical analysis will include multiple linear regression models to assess these associations. The regression models will estimate the strength and direction of the associations, controlling for covariates.
Association Between Pill Burden and Mental Health Impact in People Living With HIV | Cross-sectional assessment at baseline (one-time measurement during study enrollment).
  This outcome evaluates the association between the number of daily pills (pill burden) for HIV treatment and its impact on mental health (depression measured using the Patient Health Questionnaire-9, PHQ-9; range: 0-27, where higher scores indicate more severe depression; and anxiety measured using the Generalized Anxiety Disorder-7, GAD-7; range: 0-21, where higher scores indicate more severe anxiety). The goal is to determine whether a higher pill burden is associated with worse mental health outcomes, adjusting for potential confounding variables such as age, gender, and duration of HIV treatment. Statistical analysis will include multiple linear regression models to assess these associations. The regression models will estimate the strength and direction of the associations, controlling for covariates.
Association Between HIV Treatment Satisfaction and Stigma/Mental Health Indicators | Cross-sectional assessment at baseline (one-time measurement during study enrollment).
  This outcome evaluates the association between satisfaction with HIV treatment (measured using the HIV Treatment Satisfaction Questionnaire, HIVTSQ; range: 0-60, where higher scores indicate greater satisfaction) and indicators of stigma (HIV Stigma Scale; range: 0-48, where higher scores indicate greater stigma) and mental health (depression measured using the Patient Health Questionnaire-9, PHQ-9; range: 0-27, where higher scores indicate more severe depression; and anxiety measured using the Generalized Anxiety Disorder-7, GAD-7; range: 0-21, where higher scores indicate more severe anxiety). The goal is to determine whether higher treatment satisfaction is associated with lower levels of stigma and better mental health outcomes, adjusting for potential confounding variables such as age, gender, and duration of HIV treatment. Statistical analysis will include multiple linear regression models to assess these associations.
Assessment and comparison of HIV-Related Knowledge between Urban versus Island Settings | Cross-sectional assessment at baseline (one-time measurement during study enrollment).
  This outcome evaluates the level of knowledge about HIV using the HIV Knowledge Questionnaire-18 (HIV-KQ-18; range: 0-18, where higher scores indicate greater knowledge). The objective is to compare HIV knowledge levels between two regions and identify potential gaps. The analysis will consider key sociodemographic factors such as age, gender and education level. Statistical methods will include independent t-tests or Mann-Whitney U tests for regional comparisons, and multiple linear regression models to examine the association between knowledge scores and sociodemographic variables, adjusting for potential confounders.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saúde de Santa Maria, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No